CLINICAL TRIAL: NCT06708013
Title: The Effect of Transcranial Magnetic Stimulation Treatment on Microvasculature Stracture of the Retina and the Choroid in Treatment-Resistant Depression
Brief Title: The Effect of Transcranial Magnetic Stimulation Treatment on Microvasculature Stracture of the Retina and the Choroid
Acronym: TMS_OCT-A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Beyazit Garip, Principal Investigator, Gulhane Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 46418926/2022-334
Record Dates: First submitted 2024-10-09; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: TMS; OCTA; MACULA; RETINA; DEPRESSION
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Treatment resistant depression patient group will be evaluated before and after Transcranial Magnetic stimulation (TMS) treatment. There is a control group consist of healthy participants that will be only evaluated for ophthalmologic measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Transcranial Magnetic Stimualtion Treatment Arm (Experimental): Experimental: Treatment resistant depression group Participants will be treated with TMS using the MagVenture™ MagProX100™ device. The treatment includes 20 sessions over 4 weeks, delivering 18000 pulses in total. The stimulation targets the left dorsolateral prefrontal cortex, with parameters set to achieve optimal therapeutic effects without inducing adverse side effects. Motor threshold measurements are conducted prior to the initiation of treatment and adjusted weekly to maintain consistent treatment intensity.
  Comprehensive ophthalmologic examinations will be performed on all participants both before and after the completion of the TMS treatment. These examinations will include assessments of retinal vasculature using OCTA. The PHQ-9 and Hamilton Depression Rating Scale 17 will be conducted to evaluate changes in the severity of depressive symptoms.
  Interventions: Biological: Transcranial Magnetic Stimulation

INTERVENTIONS:
Biological: Transcranial Magnetic Stimulation — Transcranial Magnetic Stimulation Transcranial Magnetic Stimulation (TMS) is a noninvasive procedure that uses magnetic fields to stimulate nerve cells in the brain. It's primarily used to treat depression, especially in patients who haven't responded well to traditional treatments like medications or psychotherapy. The most common target is the dorsolateral prefrontal cortex, a region often underactive in people with depression. The magnetic pulses stimulate or inhibit brain activity in the targeted area. This is believed to help reset or correct patterns of neural activity associated with depression and other psychiatric disorders. TMS represents an alternative for those struggling with depression, offering a non-invasive approach with relatively few side effects and significant potential benefits

SUMMARY:
Transcranial Magnetic Stimulation (TMS) therapy is an approved and effective treatment option in treatment-resistant depression. The present study aims to investigate the effect of TMS treatment on microvasculature stracture of the retina and the choroid. These patients will be evaluated using the Optical Coherence Tomography Angiography (OCTA) device, which is quick and non-invasive, and provides volumetric data with the clinical capability of specifically localizing and delineating pathology along with the ability to show both structural and blood flow information in tandem. The main question it aims to answer is:

* Does TMS treatment influence the retinal vasculature ? The patients will visit the ophthalmology clinic before and after the TMS treatment.
* TMS treatment will be applied 5 days a week for 4 weeks.

DETAILED DESCRIPTION:
This prospective cohort study aims to investigate the impact of transcranial magnetic stimulation (TMS) on retinal microvasculature of the retina and the choroid in patients with treatment resistant depression (TRD). TRD represents a subset of major depressive disorder where patients do not adequately respond to conventional antidepressant treatments. Emerging evidence suggests that TMS, a non invasive brain stimulation technique, can effectively alleviate symptoms in TRD patients. However, the implications of TMS on ocular health, particularly the retina, remain poorly understood. This study seeks to fill this knowledge gap by assessing retinal vasculature before and after a structured TMS treatment protocol.

The study will enroll 30 patients diagnosed with TRD according to The Diagnostic and Statistical Manual of Mental Illnesses (DSM-5) criteria. Participants will undergo a TMS treatment regimen using the MagVenture™ MagProX100™ device. The treatment protocol includes 20 sessions over four weeks, delivering 18,000 pulses in total. The stimulation targets the left dorsolateral prefrontal cortex, with parameters set to achieve optimal therapeutic effects without inducing adverse side effects. Motor threshold measurements will be conducted prior to the initiation of treatment and adjusted weekly to maintain consistent treatment intensity. The control group will be consisted of 30 healthy participants. They will not be treated nor followed, they just will be evaluated for ophthalmologic measurements for once.

Comprehensive ophthalmologic examinations will be performed on all patients both before and after the completion of the TMS treatment. These examinations will include assessments of retinal vasculature using OCTA). Psychiatric assessments using the the Patient Health Questionnaire (PHQ-9) and Hamilton Depression Rating Scale (Ham17) will be conducted to evaluate changes in the severity of depressive symptoms.

The primary objective is to determine whether TMS therapy induces changes in microvasculature of the retina and the choroid in TRD patients. Secondary objectives include evaluating the safety and tolerability of TMS in this population, assessing changes in depressive symptomatology, and examining potential interactions between TMS and concurrent antidepressant use. Primary outcomes will focus on changes in retinal vasculature pre- and post TMS treatment. Secondary outcomes will assess the clinical response to TMS based on standard psychiatric scales, record any TMS-related side effects, and explore associations between treatment effects and antidepressant use.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Major Depressive Disorder according to DSM-5 TR.
* Lack of response to treatment after being administered at least two different antidepressants and anti-obsessive agents at effective doses and durations.
* The clinical condition cannot be better explained by a metabolic or organic disorder.
* Routine electroencephalography (EEG) findings before TMS do not indicate electrical activity consistent with an epileptic focus.
* Routine blood tests before TMS show no conditions that could affect treatment levels, particularly thyroid issues, vitamin deficiencies, or inflammation parameters that might cause depression or cognitive impairment (consultation with relevant departments if necessary).
* No history of hearing loss identified during routine evaluations (if a history of hearing loss exists, consultation will be requested; if none, the process will proceed accordingly).

Exclusion Criteria:

* According to the pre-TMS risk assessment form, there is a contraindication for treatment,
* Epileptic focus is detected in the pre-TMS electroencephalography findings,
* Previous head trauma, loss of consciousness and intra-cerebral surgery,
* A metal particle caused by an aneurysm clip, connection tongs or explosive substances that will affect the electromagnetic field in the brain,
* A significant disorder in the thyroid hormone profile in routine blood checks before TMS,
* A significant increase in inflammation markers in routine checks before TMS,
* A vitamin deficiency that may cause cognitive impairment or forgetfulness in routine blood checks before TMS,
* A presence of electrolyte imbalance in routine blood checks before TMS,
* The patient has previously had a psychotic attack or bipolar mood attack,
* The patient has previously had a substance-induced psychosis or bipolar mood disorder,
* The patient has previously used substances known as alcohol, drugs or stimulants according to DSM-V TR and semi-structured clinical interview (SCID-5 TR) have abuse or addiction (except if they have not used in the last 12 months or have not abused alcohol),
* Those who want to terminate TMS treatment voluntarily,
* If an unexpected clinical situation occurs during TMS treatment, the patient will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
The Effects of Transcranial Magnetic Stimulation Treatment on the Retinal Vasculature in Eyes of the Patients with Depression | From enrollment to the end of treatment at 4 weeks
  Primary Outcome Measure:
  1. The Effects of Transcranial Magnetic Stimulation Treatment on the retinal vasculature in Eyes of the Patients with TRD. The changes in the retinal vasculature in TRD patients before and after TMS treatment, as assessed by OCTA. By using OCTA, what will be measured?
  1. Capillary Density: Quantifies the density of blood vessels in the retina and choroid.
  2. Vascular Perfusion: Assesses the degree of blood flow in retinal layers.
  3. Non-Perfusion Areas: Identifies areas with reduced or absent blood flow, often indicative of ischemia or disease.
  In addition to that, Foveal Avascular Zone, Microaneurysms and Neovascularization will be assessed by using this technique. Retinal side effects related to TMS in 30 TRD patients will be evaluated using the OCTA measurement method.
The Effects of Transcranial Magnetic Stimulation Treatment on the Retinal Vasculature in Eyes of the Patients with Depression | From enrollment to the end of treatment at 4 weeks
  Primary Outcome Measure:
  Before starting TMS treatment and during the 20th session of treatment, retinal microvascular structures will be measured using OCTA. The results obtained will be compared with those of healthy controls. Changes in retinal vascular structures due to treatment and whether they differ from healthy controls will be evaluated. Another measurement involves the application of psychometric scales to TRD patients, aiming to determine the severity of the disease.
  The relationship between these two measurements will also be explored. Specifically, differences in microvascular structures before and after TMS will be examined between the group responding to treatment (achieving a 50% reduction in psychometric scale scores) and the non-responding group.
  The different measurement units obtained from these scales will be used during evaluations within and data will be integrated to provide to provide comprehensive insight.

SECONDARY OUTCOMES:
Determination of the effects of concomitant antidepressant use on retinal vascular structures using the OCTA method. | From enrollment to the end of treatment at 4 weeks
  In the treatment of TRD patients, the effectiveness, safety, and side effects of the medications used will be evaluated in detail, and it will be assessed whether the patients are using these medications at effective doses and durations. To evaluate whether these antidepressant medications have potential retinal side effects, no adjustments will be made to the patients' medication doses or the medications themselves for one month prior to TMS treatment and until the completion of 20 sessions. This approach will allow a comparison with healthy controls to determine whether the different antidepressants used have any side effects on the retina.The data collected will be combined and analyzed using advanced analytical methods to evaluate the antidepressant doses used by TRD patients undergoing TMS treatment in terms of treatment efficacy, improvement observed in psychometric scales (a reduction of more than 50% ), and their effects on retinal microvascular structures.
Determination of the effects of concomitant antidepressant use on retinal vascular structures using the OCTA method. | From enrollment to the end of treatment at 4 weeks
  To assess the effectiveness of the antidepressants administered, the HAM-17 and PHQ-9 scales will be used. A response to treatment will be defined as a 50% reduction in scores on these scales. The differences in retinal vascular structures measured by OCTA will be evaluated between the group responding to treatment and the group not responding to treatment.
  At this stage, psychometric scale data and OCTA measurements will be integrated, and advanced statistical methods will be employed to identify a retinal microvascular signature that could predict the response to TMS treatment. Additionally, it will be evaluated whether the use of specific antidepressants in conjunction with TMS has any side effects on retinal structures.
Transcranial Magnetic Stimulation Safety | From enrollment to the end of the treatment at 4 weeks.
  4. Side Effects Assessment Recording any adverse events or unexpected side effects noted during or after the TMS sessions, to evaluate the safety profile of the treatment. There is no standardized method for evaluating the side effects of TMS, a clinician will evaluate the participants for known side effects including changes in hearing, local pain, muscle contractions, headache, non-specific tingling, and discomfort.
Evaluation of the Effect of TMS Treatment on Depression Severity | From enrollment to the end of treatment at 4 weeks
  Tracking reductions in depression severity The depressive symptoms will be measured using the Patient Health Questionnaire (PHQ-9) and the Hamilton Depression Rating Scale (Ham17) before and after TMS treatment (effectiveness of the TMS protocol).
  The PHQ-9 consists of nine questions that assess symptoms of depression over the past two weeks. Each question is scored on a scale of 0 to 3, with higher scores indicating more severe symptoms. The total score ranges from 0 to 27.
  The Ham17 consists of 17 questions and it is used to determine the presence and type of depression. Each item is scored on a scale of 0 to 2, with 0 indicating no symptoms, 1 indicating mild symptoms, and 2 indicating severe symptoms. The total score ranges from 0 to 34, with higher scores indicating more severe depression.
Evaluation of the Effect of TMS Treatment on Clinical Global Impression | From enrollment to the end of treatment at 4 weeks
  The Clinical Global Impression (CGI) Scale will be used to evaluate the response of TRD patients to treatment and the improvement observed as a result of the semi-structured clinical interviews conducted. The Clinical Global Impression (CGI) Scale is a widely used tool in clinical research and practice to assess treatment outcomes in psychiatric conditions. It is simple, quick to administer, and provides a global view of a patient's condition and treatment response.
  CGI-Improvement (CGI-I):Evaluates improvement or change in the patient's condition compared to baseline.
  Rated on a 7-point scale:
  1. = Very much improved
  2. = Much improved
  3. = Minimally improved
  4. = No change
  5. = Minimally worse
  6. = Much worse
  7. = Very much worse

CONTACTS AND LOCATIONS:
Overall Officials: BEYAZIT GARİP, MD, Principal Investigator — Gulhane Training and Research Hospital
Locations (1):
- Gulhane Training and Research Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (IDP) will be shared together with the Clinical Study Report
  Supporting Information:
  * Study Protocol
  * Informed Consent Form (ICF)
  * Clinical Study Report (CSR)
Time Frame: The data will be made available immediately after the publication, and will remain available for at least 5 years.
Access Criteria: Anyone who wishes to access the data

REFERENCES:
- [Background] Genc A, Dalkiran M, Pirdogan Aydin E, Turkyilmaz Uyar E, Alkan A, Guven D, Ozer OA, Karamustafalioglu O. The alteration of retinal nerve fibre layer thickness with repetitive transcranial magnetic stimulation in patients with treatment resistant major depression. Int J Psychiatry Clin Pract. 2019 Mar;23(1):57-61. doi: 10.1080/13651501.2018.1480785. Epub 2018 Dec 31. PMID 30596524